CLINICAL TRIAL: NCT05182619
Title: Ultrasound-guided Stellate Ganglion Block Versus Nimodipine Infusion for Enhancement of Cerebral Blood Flow in Traumatic Brain Injury
Brief Title: Stellate Block Versus Nimodipine Infusion for Traumatic Brain Injury
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Khaled Mohamed Abdelaal, assistant lecturer os anesthesia and intensive care, Sohag University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: soh-Med-21-12-19
Record Dates: First submitted 2021-12-20; First posted 2022-01-10 (Actual); Last update posted 2022-01-10 (Actual); Status verified 2021-12

CONDITIONS: Traumatic Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ultrasoung guided stellate block (Active Comparator): stellate ganglion will have ultrasound-guided block via bupivacaine for sympathectomy and enhancement of cerebral blood flow
  Interventions: Procedure: ultrasound-guided stellate ganglion block
- nimodipine infusion (Active Comparator): intravenous nimodipine will be given for enhancement of cerebral blood flow
  Interventions: Procedure: ultrasound-guided stellate ganglion block

INTERVENTIONS:
Procedure: ultrasound-guided stellate ganglion block — under aseptic conditions, using the ultrasound guidance, bilateral stellate ganglion block will be done using bupivacaine and betamethasone mixture, 8 ml volume will be given for each side

SUMMARY:
the study is designed to perform an intervention for enhancement of cerebral blood flow in patients with traumatic brain injury showing vasospasm through transcranial doppler

ELIGIBILITY:
Inclusion Criteria:

* patients more than 18 ys old with isolated head trauma and traumatic brain injury

Exclusion Criteria:

* • Hemodynamic instability (mean ABP less than 70 mmHg)

  * History of severe systemic disease including cardiopulmonary failure or hepatorenal failure
  * Allergy to local anesthetics
  * Coagulation disorders
  * Abnormal neck structures disturbing normal anatomy as neck tumors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-01-01 (Estimated); Primary Completion 2023-01-01 (Estimated); Study Completion 2023-04-01 (Estimated)

PRIMARY OUTCOMES:
enhancement of cerebral blood flow | one week
  increased blood flow through middle cerebral artery and basilar artery measured by transcranial doppler ultraound

IPD SHARING:
Plan to Share IPD: Undecided